CLINICAL TRIAL: NCT06302166
Title: Effects of High Intensity Circuit Training and Intermittent Fasting on Polycystic Ovarian Syndrome
Brief Title: Effects of HICT and Intermittent Fasting on PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01720
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome; PCO
Keywords: PCO; Polycystic Ovary syndrome; Females; Body Image concerns
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity circuit training (HICT) (Active Comparator): For the group allocated with exercise, high intensity circuit training (HICT) of three supervised sessions per week for 20-30 mins will be given. HICT commenced after 10 mins low to moderate intensity warm up and after completing session ended with 10 mins cool down. Intensity of exercise will be measured on borg rating of perceived exertion (RPE). Perceived exertion is how hard you feel like your body is working. Although this is a subjective measure your exertion rating based on a 0 to 10 modified borg rating scale may provide a fairly good estimate of your actual heart rate during physical activity. 0 perceiving "no exertion at all" to 10 perceiving a "maximal exertion" of effort. A moderate intensity activity will be at 3-5 perceiving "somewhat hard", similarly 6-10 will be perceived as high intensity activity.
  Interventions: Other: High Intensity Circuit training (HICT)
- Intermittent fasting (IF) (Active Comparator): For the group allocated with intermittent fasting, a time restricted feeding (TRF) methodology will be administered. The Fasting protocol will begin with a 12-hour eating window (12:12) and will gradually go down to 8 hours eating window over a period of 8 weeks (16:8).
  Interventions: Other: Intermittent Fasting (IF)
- Combination of HICT and IF (Active Comparator): The group allocated with both exercise and intermittent fasting will be provided with both HICT for three sessions per week and 8 hours' time restricted eating.
  Interventions: Other: Combination of HICT and IF

INTERVENTIONS:
Other: High Intensity Circuit training (HICT) — High Intensity circuit training consisting of circuits of high intensity exercises and progressed up to 8 weeks will be provided.
  Arms: High Intensity circuit training (HICT)
Other: Intermittent Fasting (IF) — Time restricted feeding will be used in which the intervention will begin with a 12:12 window leading to a 16:8 IF protocol.
  Arms: Intermittent fasting (IF)
Other: Combination of HICT and IF — The participants will follow both HICT and IF for 8 weeks.
  Arms: Combination of HICT and IF

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of High intensity circuit training, Intermittent Fasting, and their combination on PCOS morphology, Anthropometrics, clinical hyperandrogenism and body image concerns in females with PCOS.

Participants will be divided into three groups who will receive High intensity circuit training, Intermittent fasting and their combination. The outcomes will be PCOS morphology, anthropometrics', clinical hyperandrogenism and body image concerns.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried females
* Diagnosed with PCOS Phenotype A based on Rotterdam Criteria:

  * PCOM on US
  * Ovulatory dysfunction
  * Clinical Hyperandrogenism (Hirsutism modified Ferriman Gallway score ≥ 8)
* Not engaged in any regular lifestyle intervention for <3 Months prior to inclusion

Exclusion Criteria:

* Use of Estrogen, Progestin or combination.
* Taking medications or supplements for Insulin resistance < 3 months prior to the inclusion
* Type I or II DM
* Hypo/hyperthyroidism
* BMI ≥27 (Obese according to BMI Asia)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
PCOS Morphology | 8th Week
  Changes from baseline PCOS morphology on the ultrasound will be done by calculating the number of follicles and measuring follicle size. For this purpose, ultrasound imaging is the best option as it is both harmless and inexpensive. PCOS is considered if on ultrasound imaging there are 12 or more than 12 follicles in the ovary and has size of 2-9 mm or volume of 10 cm 3 .

SECONDARY OUTCOMES:
Anthropometrics | 8th Week
  Changes from baseline Weight (kg) will be measured by weight scale while height (ft) will be measured by stadiometer. BMI will be calculated by dividing your weight in kilograms (kg) by your height in meters squared (m 2 ). Waist Circumference (WC) will be measured in centimeters, between the costal margin and the pelvic brim, and Hip Circumference (HC) will be measured in cm at the level of the symphysis pubis by inches tape.
Clinical Hyperandrogenism | 8th Week
  Changes from baseline Modified Ferriman Gallwey (mFG) score will be used to assess the hirsutism as a measure of clinical hyperandrogenism.
Body Image concerns | 8th Week
  Changes from baseline Body Image concerns will be measured using The BSQ which is a self-reported measurement of the body shape concerns designed for women to measure concerns about body image problems.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Bilal Hospital, Rawalpindi, Punjab Province
  - Noor Clinic, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No